CLINICAL TRIAL: NCT06625606
Title: Continuous Spinal Anesthesia for Patients Planned For Major Orthopedic Surgeries: Versus Single-Shot Spinal Anesthesia: A Case-Control Comparative Study
Brief Title: Continuous Versus Single-Shot Spinal Anesthesia for Orthopedic Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Eman M Elafifi, Lecturer of Anesthesia, Pain & ICU, Benha University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RC 5/9/2024
Record Dates: First submitted 2024-09-29; First posted 2024-10-03 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Post Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Bupivacaine

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Single-shot spinal anesthesia (SSSA) (Active Comparator): The patient's back was prepared for surgery. They were positioned on their side, with the operative side facing upward. A thin spinal needle was inserted into the L3-4 spinal interspace, after numbing the area. Once cerebrospinal fluid was confirmed, a small dose of isobaric bupivacaine was injected into the spinal canal.
  Interventions: Drug: Bupivacaine 0.5% Injectable Solution
- Continuous spinal anesthesia (CSA) (Active Comparator): A thicker needle was inserted into the L3-4 spinal interspace. After confirming cerebrospinal fluid, a thin catheter was inserted into the spinal canal and secured. An initial dose of isobaric bupivacaine was injected, followed by additional doses as needed to maintain the block height.
  Interventions: Drug: Bupivacaine 0.5% Injectable Solution
- General anesthesia (Active Comparator): General anesthesia was initiated with propofol and rocuronium. Anesthesia was maintained with isoflurane, with additional rocuronium and fentanyl as needed. Breathing was controlled by the ventilator, and muscle relaxation was reversed at the end of surgery.
  Interventions: Drug: Isoflurane Inhalant Product

INTERVENTIONS:
Drug: Bupivacaine 0.5% Injectable Solution — The patient's back was prepared for surgery. They were positioned on their side, with the operative side facing upward. The L3-4 spinal interspace was identified, and numbed, and a thin spinal needle was inserted. After confirming Cerebrospinal Fluid (CSF), 12.5 mg of isobaric bupivacaine 0.5% was injected into the spinal canal.
  Arms: Single-shot spinal anesthesia (SSSA)
Drug: Bupivacaine 0.5% Injectable Solution — The L3-4 spinal interspace was identified, numbed, and a thicker needle (Tuohy needle) was inserted. After confirming Cerebrospinal Fluid (CSF), a thin catheter was inserted into the spinal canal and secured. An initial dose of 1 ml isobaric bupivacaine 0.5% was injected, followed by additional doses as needed to maintain the block height.
  Arms: Continuous spinal anesthesia (CSA)
Drug: Isoflurane Inhalant Product — General anesthesia was initiated with propofol and rocuronium. Anesthesia was maintained with isoflurane, with additional rocuronium and fentanyl as needed. Breathing was controlled by the ventilator, and muscle relaxation was reversed at the end of surgery.
  Arms: General anesthesia

SUMMARY:
A study was conducted to compare the effectiveness of continuous spinal anesthesia (CSA), single-shot spinal anesthesia (SSSA), and general anesthesia (GA) in patients over 60 years of age undergoing elective surgical repair of a fractured neck of femur. One hundred and five patients were randomly assigned to one of the three groups. The SSSA group received a single intrathecal injection of isobaric bupivacaine 0.5%, while the CSA group received multiple injections of the same anesthetic through a catheter placed in the subarachnoid space. The GA group received isoflurane anesthesia. Intraoperatively, blood pressure was monitored to assess the frequency of hypotension and the required dose of ephedrine. Additionally, the total dose of bupivacaine administered and the frequency of intraoperative fentanyl were recorded. Postoperatively, the duration of postoperative analgesia, pain scores, and need for additional pain medication were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) grade ≤III;
* Patients were assigned for elective surgical intervention for Fixation of Neck Femur;
* Patients were free of exclusion criteria.

Exclusion Criteria:

* Patients of American Society of Anesthesiologists (ASA) grade >III;
* Patients who had uncontrolled hypertension and/or diabetes mellitus;
* Patients who had uncompensated cardiac, renal, or hepatic diseases;
* Patients with coagulopathy, spinal deformity, allergy, or contraindication for the used drugs;
* Patients who refused to sign the informed consent were excluded from the study.

Ages: 60 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2024-11-15 (Actual); Study Completion 2024-12-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients reporting at least a 50% reduction in pain (measured by Numerical Rating Scale) post orthopedic surgery. | 3 months
  Value of Continuous Spinal Anesthesia in Pain Reduction Post-operative manifested by Total dose of Post Operative analgesia.

CONTACTS AND LOCATIONS:
Locations (1):
- Benha University, Banhā, El Qalyoubia, Egypt